CLINICAL TRIAL: NCT04421768
Title: Effects of Systematic Cervical Exam Training on Labor and Delivery Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00064273
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-06

CONDITIONS: Delivery Problem; Cervix; Pregnancy; Pregnancy Related
Keywords: vaginal delivery; labor cervical exam; labor and delivery
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Intervention Model Description: The total number of exams per hour of labor or triage stay and exam discrepancy between 2 examiners will be compared between the 6 month time period before training and 6 months after all nurses have completed the training
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- systematic cervical exam training--retrospective measures (Experimental): Effects of systematic cervical exam training on Labor and Delivery Care The total number of exams per hour of labor or triage stay and exam discrepancy between 2 examiners who performed exams less than 30 minutes apart will be compared between the 6 month time period before the unit wide training and 6 months after completing training
  Interventions: Behavioral: cervical exam training
- systematic cervical exam training--prospective measures (Experimental): Effects of systematic cervical exam training on Labor and Delivery care Patient will be approached to obtain consent for them to have 2 cervical exams performed one after the other when an exam is clinically indicated. The discrepancy between the 2 examiners will be compared between the 6 month time period before the unit wide training and 6 months after completion of the training.
  Interventions: Behavioral: cervical exam training

INTERVENTIONS:
Behavioral: cervical exam training — Each nurse will then examine 1 sets of 10 high-fidelity silicone task trainers approximately three per week for a maximum of 20 sessions (200 repetitions total). For each set of 10 exams, the estimates will recorded on an answer sheet. A cumulative summation analysis will be performed on each participant. When an individual nurse achieves competence her training will be suspended

SUMMARY:
All physicians, nurses, and nurse midwives working on Labor and Delivery will be required to complete cervical exam simulation training. Data before and after institution of the training will be compared to determine if the training leads to less cervical exams during labor and increases consistency between examiners

DETAILED DESCRIPTION:
The labor cervical exam is the cornerstone of the management of labor as the accurate assessment of cervical dilation and effacement are crucial in recognizing a normal labor from and abnormal one. To enhance accuracy and precision among healthcare providers working on Labor and Delivery we have created a high fidelity cervical exam simulator. All providers working on Labor and Delivery Repetitive will be required to practice on the simulators until a pre-specified level or accuracy is achieved. We will prospectively and retrospectively assess the number of cervical exams a women receives and the discrepancy between exams performed by 2 different providers both before and after the training is instituted.

ELIGIBILITY:
Inclusion Criteria:

Healthcare providers:

• physicians, midwives, and labor and delivery nurses working on the Labor and Delivery unit within the Wake Forest Baptist Birth Center

Patients:

• any pregnant women receiving care on the Labor and Delivery unit of Wake Forest Baptist Birth Center

Exclusion Criteria:

Healthcare providers:

• none

Patients:

* placenta previa
* vasa previa
* any other contraindication to cervical exam

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Physicians, nurses and nurse midwives: any gender Patients: pregnant women only
Enrollment: 1125 (Estimated)
Dates: Start 2020-07-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of repetitions needed to obtain competence | 3 month training period
  The number of simulated cervical exams each provider needs to reach a pre-specified level of accuracy.
Number of exams patients receive | Six months period before training
  Number of exams per hour of labor or triage visit
Number of exams patients receive | Six month post training
  Number of exams per hour of labor or triage visit

SECONDARY OUTCOMES:
Discrepancy between 2 cervical exam assessments--retrospective | Six months period before training and Six months period post training completion
  Discrepancy between 2 exam assessments performed less than 30 minutes apart by 2 different examiners:
  Cervix Dilation will be reported as 1-10 cm Cervix Effacement will be reported as 0% -100%
Discrepancy between 2 cervical exam assessments--prospective | Six months period before training and Six months period post training completion
  Discrepancy between 2 exam assessments performed one after the other by 2 different examiners:
  Cervix Dilation will be reported as 1-10 cm Cervix Effacement will be reported as 0% -100%

CONTACTS AND LOCATIONS:
Overall Officials: Joshua F Nitsche, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States